CLINICAL TRIAL: NCT03872570
Title: Comparison of the Hemodynamic Effects of Phenylephrine and Norepinephrine in Patients Undergoing Deep Inferior Epigastric Perforator (DIEP) Flap Surgery.
Brief Title: Effect of Phenylephrine Versus Norepinephrine on Venous Return
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Dr. Alain Kalmar, MD, PhD, Staff Anesthesist, Algemeen Ziekenhuis Maria Middelares
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MMS.2019.008
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Arterial Hypotension
Keywords: cardiac output; pulse pressure variation; fluid responsiveness; hemodynamic monitoring
MeSH Terms: conditions — Hypotension | interventions — Phenylephrine; Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- phenylephrine (Active Comparator): starts at 15 µg/kg/h phenylephrine and titrated to main a minimal systolic blood pressure of 100 mmHg
  Interventions: Drug: Phenylephrine
- norepinephrine (Active Comparator): starts at 1.5 µg/kg/h phenylephrine and titrated to main a minimal systolic blood pressure of 100 mmHg
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Phenylephrine — intravenous administration
  Arms: phenylephrine
Drug: Norepinephrine — intravenous administration
  Arms: norepinephrine

SUMMARY:
Induction of general anesthesia often induces a decrease in the mean arterial blood pressure (MAP) caused by arterial and venous dilatation. Fluid administration is conventionally used to increase the patient's total blood volume, but is often associated with multiple adverse events such as postoperative edema.

Arterial hypotension can also be treated by vasopressor agents such as norepinephrine and phenylephrine which mainly increase the blood pressure by arterial vasoconstriction.

Compared to phenylephrine, norepinephrine has a shorter half-life (2 - 3 minutes) and improves the MAP by increase in cardiac contractility. In a recent study at our department it was demonstrated that besides arterial vasoconstriction, phenylephrine also improves venous return and cardiac output by venous vasoconstriction.

The aim of this study is to compare the hemodynamic effects of both vasopressor agents in patients undergoing deep inferior epigastric perforators (DIEP) flap surgery. If significant differences between both agents are demonstrated, these findings can provide an important basis for future recommendations.

DETAILED DESCRIPTION:
In consecutive patients scheduled for DIEP flap surgery, all hemodynamic and respiratory variables are recorded electronically for subsequent off line analysis.

A systolic blood pressure of minimal 100 mmHg will be maintained during surgery by optimization of the cardiac preload and titrated norepinephrine (1.5 µg/kg/h) or phenylephrine (15 µg/kg/h) administration. Cardiac preload optimization will be based on pulse pressure variation (PPV) measurement, which is calculated by pulse contour analysis of the radial arterial pressure curve. Following the international goal-directed fluid therapy guidelines, plasmalyte will be administrated if the PPV>11%.

The tricuspid annular plane systolic excursion (TAPSE) will be measured by transthoracic echocardiography (TTE) to evaluate the inotropic effect of norepinephrine and phenylephrine. In addition, TTE will be used to measure the cardiac output to calibrate the PPV measurements.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* patients scheduled for DIEP flap surgery

Exclusion Criteria:

* unwilling or unable to grant written informed consent
* contra-indications for phenylephrine or norepinephrine
* cardiac arrhythmia
* no necessity for pharmacological blood pressure management

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
pulse pressure variation | perioperative
  the evolution of the pulse pressure variation in a time course of 20 minutes after the start of phenylephrine/norepinephrine administration

SECONDARY OUTCOMES:
mean arterial blood pressure | perioperative
  the evolution of the mean arterial blood pressure in a time course of 20 minutes after the start of phenylephrine/norepinephrine administration
cardiac output | perioperative
  the evolution of the cardiac output in a time course of 20 minutes after the start of phenylephrine/norepinephrine administration
stroke volume (variation) | perioperative
  the evolution of the stroke volume (variation) in a time course of 20 minutes after the start of phenylephrine/norepinephrine administration
heart rate | perioperative
  the evolution of the heart rate in a time course of 20 minutes after the start of phenylephrine/norepinephrine administration
ventilation frequency | perioperative
  the evolution of the ventilation frequency in a time course of 20 minutes after the start of phenylephrine/norepinephrine administration
end-tidal CO2 | perioperative
  the evolution of the end-tidal CO2 in a time course of 20 minutes after the start of phenylephrine/norepinephrine administration
tidal volume | perioperative
  the evolution of the tidal volume in a time course of 20 minutes after the start of phenylephrine/norepinephrine administration
TAPSE | perioperative
  the evolution of the tricuspid annular plane systolic excursion in a time course of 20 minutes after the start of phenylephrine/norepinephrine administration

CONTACTS AND LOCATIONS:
Overall Officials: Alain F Kalmar, MD, PhD, Principal Investigator — Maria Middelares Hospital
Locations (1):
- General Hospital Maria Middelares, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalmar AF, Allaert S, Pletinckx P, Maes JW, Heerman J, Vos JJ, Struys MMRF, Scheeren TWL. Phenylephrine increases cardiac output by raising cardiac preload in patients with anesthesia induced hypotension. J Clin Monit Comput. 2018 Dec;32(6):969-976. doi: 10.1007/s10877-018-0126-3. Epub 2018 Mar 22. PMID 29569112
- [Background] O'Connell TD, Jensen BC, Baker AJ, Simpson PC. Cardiac alpha1-adrenergic receptors: novel aspects of expression, signaling mechanisms, physiologic function, and clinical importance. Pharmacol Rev. 2013 Dec 24;66(1):308-33. doi: 10.1124/pr.112.007203. Print 2014. PMID 24368739
- [Background] Beloeil H, Mazoit JX, Benhamou D, Duranteau J. Norepinephrine kinetics and dynamics in septic shock and trauma patients. Br J Anaesth. 2005 Dec;95(6):782-8. doi: 10.1093/bja/aei259. Epub 2005 Oct 14. PMID 16227334
- [Background] Hengstmann JH, Goronzy J. Pharmacokinetics of 3H-phenylephrine in man. Eur J Clin Pharmacol. 1982;21(4):335-41. doi: 10.1007/BF00637623. PMID 7056280